CLINICAL TRIAL: NCT07202052
Title: A Randomised Platform Trial Evaluating the Role of Interventions to Prevent Infection in Patients With Acquired Hypogammaglobulinemia Secondary to Haematological Malignancies - RATIONAL-PT (Core)
Brief Title: Role of Antibiotic Therapy or Immunoglobulin On iNfections in hAematoLogy Platform Trial (RATIONAL-PT)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRU-RPT-22; TRU-RPT-22 (Other: Monash University)
Record Dates: First submitted 2025-09-24; First posted 2025-10-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Myeloma; Non-Hodgkin's Lymphoma; Leukemia
Keywords: immunoglobulin; antibiotics; myeloma; leukaemia; lymphoma; non Hodgkins; infection; infections; blood; cancer; haematology
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma, Non-Hodgkin; Leukemia; Lymphoma; Infections; Neoplasms | interventions — Immunoglobulins, Intravenous; Trimethoprim, Sulfamethoxazole Drug Combination; Amoxicillin-Potassium Clavulanate Combination; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Up to 900 participants will be recruited to the RATIONAL-PT, including up to 300 per domain. The aim of the platform is to determine optimal supportive care interventions for patients with haematological malignancies. The primary outcome for the platform is Event-free survival (EFS), defined as time from randomisation (or, in domains with a single treatment arm, time from registration) until occurrence of a Grade 3 or higher infection (as defined by CTCAE Version 5), or death from any cause. Data from each domain will contribute to the primary analysis.
Masking Description: An independent outcome adjudication committee will meet to review and adjudicate infection outcome data. These committee members will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Start Immunoglobulin (Other): Patients eligible to start immunoglobulin are randomly assigned to:
  * receive either prophylactic antibiotic
  * or Ig replacement.
  Interventions: Biological: Intravenous immunoglobulin; Drug: Trimethoprim / Sulfamethoxazole
- Stop Immunoglobulin (Other): Patients eligible to stop immunoglobulin are randomly assigned to:
  * Stop Ig and take daily antibiotics
  * Stop Ig and take antibiotics only when infections occur
  * Continue Ig therapy
  Interventions: Biological: Intravenous immunoglobulin; Drug: Trimethoprim / Sulfamethoxazole; Drug: Amoxicillin clavulanic acid
- Dose Immunoglobulin (Other): Patients receiving IVIg are randomly assigned to:
  * Continue with standard dose (0.4 g/kg)
  * Switch to a lower dose (0.25 g/kg)
  Interventions: Biological: Intravenous immunoglobulin (IVIG)

INTERVENTIONS:
Biological: Intravenous immunoglobulin — (IVIg) intravenous immunoglobulin every 4 weeks ± 1 week at a dose of 0.4g/kg, modified to achieve an (IgG) immunoglobulin G trough level of at least lower limit of age-specific serum IgG reference range; or SCIg, weekly, may be used in patients who meet local criteria for home-based self-administration in centres with established SCIg programs. Dosing is usually given at 100mg/kg/week, modified to achieve an IgG steady state level of at least the lower limit of the serum reference range. A loading IVIg dose may be given in the first month if required.
  Other Names: Subcutaneous immunoglobulin
  Arms: Start Immunoglobulin; Stop Immunoglobulin
Drug: Trimethoprim / Sulfamethoxazole — Once daily trimethoprim-sulfamethoxazole (co-trimoxazole) 160mg/800mg. Doxycycline 100mg daily as an alternative for patients with hypersensitivity to co-trimoxazole.
  Other Names: co-trimoxazole
  Arms: Start Immunoglobulin; Stop Immunoglobulin
Drug: Amoxicillin clavulanic acid — Patients will be provided with amoxycillin/clavulanic acid 1750-2000mg/250mg and ciprofloxacin 750 mg to keep at home for initial use if symptoms of infection develop, with immediate review by their treating clinical team, or nearest emergency department or medical practitioner with phone contact to treating team if most practical. Clindamycin 600 mg is permitted as an alternative to amoxycillin/clavulanic acid for patients with hypersensitivity to penicillin. Ciprofloxacin is omitted for participants with hypersensitivity.
  Other Names: Ciprofloxacin
  Arms: Stop Immunoglobulin
Biological: Intravenous immunoglobulin (IVIG) — Arm A: Low dose (IgRT) immunoglobulin replacement therapy: Participants will be treated with intravenous immunoglobulin monthly (every 4 weeks ± 1 week) at a dose of 0.25g/kg. No dose adjustment for trough serum IgG levels is required.
  Arm B: Usual dose: Participants will be treated with intravenous immunoglobulin monthly (every 4 weeks ± 1 week) at a dose of 0.4g/kg, modified to achieve an IgG trough level of at least lower limit of age-specific serum IgG reference range.
  Arms: Dose Immunoglobulin

SUMMARY:
This is an adaptive platform study to find out how safe and effective different strategies are in comparison to each other, for preventing infection in patients with blood cancers.

It is a comparison between Immunoglobulin and antibiotics use.

DETAILED DESCRIPTION:
This study is being conducted to find out how safe and effective different strategies of infection prevention are in comparison to each other, for preventing infection in patients with blood cancers. The best way to find out this information is to directly compare the effect of different treatment strategies in patients with blood cancers. We want to know how these different treatments impact on your health and your use of healthcare services.

This research project uses an Adaptive Platform Design. This design allows the researchers to compare multiple infection prevention strategies within the same trial at the same time (rather than running separate trials), to analyse results as the trial occurs and to add new research questions during the course of the trial.

The treatments that you may receive as part of the study will be determined by which domain(s) of the platform you participate in. By combining data collected within each domain as part of the platform, the researchers can investigate and compare treatment strategies and infection outcomes across a broader range of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than or equal to 18 years of age
2. Diagnosis of haematological malignancy, including (CLL) chronic lymphocytic leukemia, (MM) multiple myeloma or (NHL) non-Hodgkin's lymphoma.
3. Eligible to receive or currently receiving Ig (IV or subcutaneous - SCIg) replacement for history of recurrent or severe infection(s) and IgG less than the lower limit of the reference range (excluding paraprotein) OR IgG<4g/L (excluding paraprotein)
4. Life expectancy > 12 months
5. Able to give informed consent

Exclusion Criteria:

1. Treating team deems enrolment in the study is not in the best interests of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Defined as time from randomisation (or, in domains with a single treatment arm, time from registration) until occurrence of a Grade 3 or higher infection (as defined by CTCAE Version 5), or death from any cause.

SECONDARY OUTCOMES:
Occurrence of at least one Grade 3 or higher infection(s) from randomisation to 12 months | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Occurrence of at least one Grade 3 or higher infection(s) from randomisation to 12 months
Occurrence of one or more clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Occurrence of one or more clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) from randomisation to 12 months.
Number of clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Number of clinically documented infections (symptoms/signs of infection requiring antimicrobial treatment) from randomisation to 12 months.
Occurrence of one or more microbiologically documented infections from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Occurrence of one or more microbiologically documented infections from randomisation to 12 months.
Number of microbiologically documented infections from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Number of microbiologically documented infections from randomisation to 12 months.
All-cause mortality at 12 months | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  All-cause mortality at 12 months
Infection-related mortality at 12 months | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Infection-related mortality at 12 months
Time free from hospitalisation with antimicrobial administration with therapeutic intent from randomisation to 12 months. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Time free from hospitalisation with antimicrobial administration with therapeutic intent from randomisation to 12 months.
Occurrence of one or more treatment-related adverse events | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  An adverse event includes any untoward medical occurrence that is not necessarily caused by the trial treatment. Examples of adverse events might include symptoms such as nausea, diarrhoea or headache.
  Adverse events will be collected via clinical examination, hospital medical record, or self-report to study team or via study diary. Adverse events will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5. Relationship to treatment will be assessed by an Investigator at the trial site.
Number of treatment-related adverse events. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  An adverse event includes any untoward medical occurrence that is not necessarily caused by the trial treatment. Examples of adverse events might include symptoms such as nausea, diarrhoea or headache.
  Adverse events will be collected via clinical examination, hospital medical record, or self-report to study team or via study diary. Adverse events will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5. Relationship to treatment will be assessed by an Investigator at the trial site.
Isolation of fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms from randomisation to 12 months | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Isolation of fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms from randomisation to 12 months
Number of infections with fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms isolated from randomisation to 12 months | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Number of infections with fluoroquinolone resistant organisms, co-trimoxazole resistant organisms, extended spectrum beta lactamases or multidrug resistant organisms isolated from randomisation to 12 months
Quality of Life (QoL) measured at randomisation then 3, 6, 9 and 12 months, using the questionnaire. | Randomisation, Month 3, Month 6, Month 9 and Month 12
  Quality of Life (QoL) measured at randomisation then 3, 6, 9 and 12 months, using the questionnaire.
Costs associated with allocated treatment arm and infections during study. | 12 months following randomisation (or, in domains with a single treatment arm, time from registration)
  Costs of infections and trial interventions will be estimated based on trial treatment and adverse event data within the hospital medical record, as well as linked data obtained from the Medicare Benefits Scheme (MBS), Pharmaceutical Benefits Scheme (PBS) and Australian Immunisation Register (AIR). Data from the quality of life questionnaires will be used to calculate quality adjusted life years.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe McQuilten, Professor, Principal Investigator — Monash University
Locations (3):
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Hospital, Melbourne, Victoria
  - Northern Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly available. Data will only be presented as a whole, no individual data will be published or presented.

REFERENCES:
- See also: Study Website — https://rationaltrial.com

DOCUMENTS (1):
  • Study Protocol (2023-11-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT07202052/Prot_000.pdf